CLINICAL TRIAL: NCT06640842
Title: Brain Health in Midlife (ADORE BRAIN)
Brief Title: Brain Health in Midlife
Acronym: ADORE BRAIN
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00160885; P30AG072973 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-10-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Brain Health; Gestational Hypertension; Alzheimer Disease; Dementia; Cardiovascular Diseases; Pregnancy Related; Pre-Eclampsia
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Alzheimer Disease; Dementia; Cardiovascular Diseases; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertensive disorder of pregnancy: Women who were diagnosed with a hypertensive disorder of pregnancy during the ADORE study participation.
  Interventions: Diagnostic Test: A combination of various test and biomarkers will be completed to understand the effect of hypertensive disorders of pregnancy in brain health in midlife.
- Healthy pregnancy: Women who participated in the ADORE study and had a healthy pregnancy during their participation.
  Interventions: Diagnostic Test: A combination of various test and biomarkers will be completed to understand the effect of hypertensive disorders of pregnancy in brain health in midlife.

INTERVENTIONS:
Diagnostic Test: A combination of various test and biomarkers will be completed to understand the effect of hypertensive disorders of pregnancy in brain health in midlife. — Participants will be asked to complete a blood draw, 5-lead ECG, MRI, a series of cognitive assessments, dietary assessments, monitor sleep and physical activity and DXA scan.

SUMMARY:
The purpose of this study is to learn if hypertensive disorders during pregnancy affects brain health in midlife.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the ADORE trial ( R01 HD083292)

Exclusion Criteria:

* History of seizures or Epilepsy
* Pregnant at screening
* Ineligible to complete MRI due to metal in the body

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who previously participated in the ADORE, received a hypertensive disorder diagnosis or had a healthy pregnancy during their participation.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic markers of middle age women | Baseline
  Assess cardiometabolic marker values differences between the women diagnosed with a hypertensive disorder of pregnancy to the values of the healthy control.
Neurovascular hemodynamics of middle age women | Baseline
  Assess differences in heart rate via an ECG, and beat to beat blood pressure, cerebral blood flow, and pulse wave velocity) between the women diagnosed with hypertensive disorder of pregnancy to the values of the healthy control.
Brain structure & function of middle age women | Baseline
  Assess differences in MRI MPRAGE, fMRI and DTI sequencing scan between the women diagnosed with hypertensive disorder of pregnancy to the values of the healthy control.
Alzheimer's disease-related plasma biomarkers of middle age women | Baseline
  Assess value differences in a predetermined Alzheimer's disease-related plasma biomarkers between the women diagnosed with hypertensive disorder of pregnancy to the values of the healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Holly R Hull, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided